CLINICAL TRIAL: NCT03936946
Title: The 28 Day Challenge
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources not secured
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Snyder, Chairman and Professor of Genetics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50298
Record Dates: First submitted 2019-04-15; First posted 2019-05-03 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Depression; Anxiety; Stress; Hope
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to Group 1, Group 2, or Group 3. Group 1 begins the 28 day challenge in October (while group 2 acts as a passive control) and Group 2 begins the 28 day challenge 1 months late (while Group 1 receives no further intervention). Group 3 will begin the 28 day challenge concurrent with Group 1, but will listen to different audio clips than Group 1 (blinded).
Who Masked: Participant
Masking Description: Participants will not be told what the intervention is until they are assigned (i.e. each group will not know what they will be listening to ahead of time or what other groups are listening to).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1--October Start Audio Content 1 (Experimental): This group will listen to audio content 1 daily for 28 days beginning in October, and then will receive no further intervention
  Interventions: Behavioral: Audio Content 1
- Group 2--November Start Audio Content 1 (Other): This group will not be assigned to any interventions during the first month of the trial and will act as a passive control group at that time. They will be assigned to listen to audio content 1 daily for 28 days beginning in November.
  Interventions: Behavioral: Audio Content 1
- Group 3--October Start Audio Content 2 (Sham Comparator): This group will listen to audio content 2 daily for 28 days beginning in October, and then will receive no further intervention.
  Interventions: Behavioral: Audio Content 2

INTERVENTIONS:
Behavioral: Audio Content 1 — ~30 minute daily audio recordings of content 1 for 28 days
  Arms: Group 1--October Start Audio Content 1; Group 2--November Start Audio Content 1
Behavioral: Audio Content 2 — ~30 minute daily audio recordings of content 2 for 28 days
  Arms: Group 3--October Start Audio Content 2

SUMMARY:
The purpose of this study is to determine how a 28 Day Challenge influences mental health and well-being. This is a blinded study. Participants both with and without depression and anxiety, will be included. A moderation analysis will be performed to see whether changes in depression after the intervention are a function of baseline depression and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* English Fluency

Exclusion Criteria:

* Severe hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-10 (Estimated); Primary Completion 2020-07-10 (Estimated); Study Completion 2020-10-10 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Heath Questionnaire-9 (PHQ-9) | Baseline, 1 months
  The PHQ-9 is a self-administered survey used for diagnosing depression and assessing depression severity. It measures each of the 9 DSM-IV/V diagnostic criteria for depression on a 0-3 scale. Depression Severity is measured as follows: 0 none, 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Validity has been assessed against structured clinical interviews. PHQ-9 scores ≥10 exhibited a sensitivity of 88% and a specificity of 88% for major depression.
  DSM = The Diagnostic and Statistical Manual of Mental Disorders
Change in Patient Heath Questionnaire-9 (PHQ-9) | Baseline, 3 months
  The PHQ-9 is a self-administered survey used for diagnosing depression and assessing depression severity. It measures each of the 9 DSM-IV/V diagnostic criteria for depression on a 0-3 scale. Depression Severity is measured as follows: 0 none, 1-4 minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Validity has been assessed against structured clinical interviews. PHQ-9 scores ≥10 exhibited a sensitivity of 88% and a specificity of 88% for major depression.
  DSM = The Diagnostic and Statistical Manual of Mental Disorders
Change in Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 1 months
  The GAD-7 is a self report-based survey that assesses generalized anxiety disorder and severity on a 7-item scale. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. The GAD-7 was compared to diagnoses by mental health professionals. Using scores >/= 10, It has sensitivity of 89% and specificity of 82%.
Change in Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 3 months
  The GAD-7 is a self report-based survey that assesses generalized anxiety disorder and severity on a 7-item scale. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. The GAD-7 was compared to diagnoses by mental health professionals. Using scores >/= 10, It has sensitivity of 89% and specificity of 82%.
Change in Perceived Stress Scale-10 (PSS-10) | Baseline, 1 months
  The Perceived Stress Scale-10 (PSS-10) measures global perceived stress via self-report on a ten item scale. Scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Total scores ranging from 0-13 would be considered low stress. Total scores ranging from 14-26 would be considered moderate stress. Total scores ranging from 27-40 would be considered high perceived stress.
Change in Perceived Stress Scale-10 (PSS-10) | Baseline, 3 months
  The Perceived Stress Scale-10 (PSS-10) measures global perceived stress via self-report on a ten item scale. Scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Total scores ranging from 0-13 would be considered low stress. Total scores ranging from 14-26 would be considered moderate stress. Total scores ranging from 27-40 would be considered high perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Michasel Snyder, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data